CLINICAL TRIAL: NCT04911244
Title: Assessment of Different Diagnostic Modalities for Detection of Ventilator Associated Pneumonia
Brief Title: Diagnostic Modalities for VAP Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Refaat Mahmoud, Principle investigator, Assiut University
Allocation: Non-Randomized | Model: Single Group | Purpose: Diagnostic
Other Study IDs: VAP diagnosis
Record Dates: First submitted 2021-05-24; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAP group (Experimental): patients confirmed diagnosis of VAP with bronchoalveolar lavage
  Interventions: Diagnostic Test: bronchoalveolar lavage
- Non VAP group (Experimental): patients confirmed not VAP with bronchoalveolar lavage
  Interventions: Diagnostic Test: bronchoalveolar lavage

INTERVENTIONS:
Diagnostic Test: bronchoalveolar lavage — endobronchial sampling through bronchoscopy
  Other Names: protected endotracheal aspirate

SUMMARY:
asses diagnostic performance of different methods for detection of ventilator associated pneumonia.

DETAILED DESCRIPTION:
Ventilator associated pneumonia (VAP) is a common cause of nosocomial infection, that can complicate mechanical ventilation and is related to significant utilization of health-care resources.

The diagnosis of VAP is subjected to considerable interobserver variability. The Centers for Disease Control and Prevention (CDC) definition of VAP uses a combination of clinical, radiographic, and micro-biological criteria for diagnosis, but in the absence of a definite diagnostic test, the accurate diagnosis and treatment of VAP is limited.

The clinical pulmonary infection score (CPIS) was developed to objectively diagnose VAP and assign points on the basis of clinical and radiographic data, but its role in diagnosing pneumonia remains controversial .

Lung ultrasound (LUS) is a simple, non irradiating, noninvasive, cost-effective, bedside technique. It has been successfully applied for monitoring aeration and monitoring antibiotic efficacy in ventilator-associated pneumonia (VAP). However, no scientific evidence is yet available on whether LUS reliably improves the diagnosis of VAP.

Quantitative bacterial cultures of the specimen obtained from the lower airways using bronchoscope were proposed for VAP diagnosis with a cut off value of 104 colony-forming unit/ml. However, microbiological cultures cannot guide the early clinical management of patients with a suspected VAP, as they need at least 24 hours for preliminary results. So, starting antibiotics remains a challenge. Moreover, bronchoscopy is not always easy to perform in hypoxemic patients and not promptly available in all ICUs. Therefore, it can be replaced by tracheal aspirate microbiological samples.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients mechanically ventilated for at least 48 hours in Respiratory ICU were included in the study.

who had:

* Clinically suspected VAP according to simplified Clinical Pulmonary Infectious Score exceeding 6.
* Or new or extension of a radiological image with at least two of the following clinical criteria:

  * Body temperature ≥ 38.5 ° C or <36 ° C.
  * Leukocytes> 10 * 103 / ml or <4 * 103/ ml or > 10% immature cells (in the absence of other known causes).
  * Purulent tracheal secretions.
  * Hypoxemia with PaO2 <60 mmHg or a PaO2 / FiO2 <300.

Exclusion Criteria:

* Patients with diagnosis of community acquired pneumonia or hospital acquired pneumonia before starting of mechanical ventilation.
* Patients who are contraindicated for bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
To detected diagnostic accuracy of chest ultrasound in VAP. | 3 years
  To identify sensitivity and specificity of chest ultrasound in VAP diagnosis
To detected diagnostic accuracy of protected endotracheal aspirate in VAP. | 3 years
  To identify sensitivity and specificity of protected endotracheal aspirate in VAP diagnosis
To detected diagnostic accuracy of usual endotracheal aspirate in VAP. | 3 years
  To identify sensitivity and specificity of usual endotracheal aspirate in VAP diagnosis
To detected diagnostic accuracy of chest X-ray in VAP. | 3 years
  To identify sensitivity and specificity of chest X-ray in VAP diagnosis

REFERENCES:
- [Background] Nair GB, Niederman MS. Ventilator-associated pneumonia: present understanding and ongoing debates. Intensive Care Med. 2015 Jan;41(1):34-48. doi: 10.1007/s00134-014-3564-5. Epub 2014 Nov 27. PMID 25427866
- [Background] Bouhemad B, Liu ZH, Arbelot C, Zhang M, Ferarri F, Le-Guen M, Girard M, Lu Q, Rouby JJ. Ultrasound assessment of antibiotic-induced pulmonary reaeration in ventilator-associated pneumonia. Crit Care Med. 2010 Jan;38(1):84-92. doi: 10.1097/CCM.0b013e3181b08cdb. PMID 19633538
- [Background] Mongodi S, Via G, Girard M, Rouquette I, Misset B, Braschi A, Mojoli F, Bouhemad B. Lung Ultrasound for Early Diagnosis of Ventilator-Associated Pneumonia. Chest. 2016 Apr;149(4):969-80. doi: 10.1016/j.chest.2015.12.012. Epub 2015 Dec 22. PMID 26836896